CLINICAL TRIAL: NCT03402256
Title: Text Messaging to Reduce Alcohol Relapse in Liver Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1210011022
Record Dates: First submitted 2017-12-13; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Alcoholic Liver Disease
Keywords: Mobile Technology; Alcohol; Alcoholic Liver Disease; Ethyl Glucuronide
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the Text Message intervention or to Standard Care based on a preset randomization schedule generated via computer by a statistician.
Who Masked: Care Provider
Masking Description: All clinical members of the liver transplantation service will be blind to the results of self-report data collected during the study and to urine toxicology results. The PI and Co-I, who also serves as the Project Manager, will not be blind to participant condition. The Research Assistant will not be blind to the participant condition after delivery of the study-provided cell phone to participants randomized to the Text Message condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message (TM) (Experimental): Participants will receive daily text messages and all elements of standard care. They received 3 text messages per day for the first four weeks of the study and 3 messages per week for the last four weeks. Key domains of message topics were chosen based on the content of evidence-based, relapse prevention treatment. Daily messages determined current level of functioning and provide intervention messages in response. Text messages will be sent via Google Voice on a research computer. Participants will respond to the text messages either with a specified response (e.g. YES/NO) or a generic response (e.g. "1"). Some messages will ask for a specific reply in response to a question. Based on the participant's response (e.g. "high," "med," "low"), the research assistant will respond with a text message tailored to the participant's message. All text messages will be sent to the HIC in an amendment to this protocol for approval.
  Interventions: Behavioral: Text Message
- Standard Care (SC) (No Intervention): Participants will receive only standard care provided by the liver transplantation team. No additional behavioral or psychosocial interventions will be provided. All aspects of care received by SC participants will also provided to the TM condition participants. Medical care will be managed by medical specialty providers. SC condition participants will receive behavioral treatment within the liver transplantation clinic by psychology fellows and/or psychologists/psychiatrists. Treatment schedules and session topics will be determined by individual providers, per usual practice.
  These participants will receive only study-specific assessments. Participants in this condition will complete assessments at baseline, 4-weeks and 8-weeks that measure self- reported substance use, stress, and coping skills. At each in-person assessment, participants will provide urine for EtG analysis and will be compensated.

INTERVENTIONS:
Behavioral: Text Message — In addition to the SC interventions, participants in the Text Message condition received text messages. Participants received 3 text messages per day for the first four weeks of the study and 3 messages per week for the last four weeks. Participants will receive messages targeting known predictors of alcohol abstinence and relapse, including (1) craving, (2) identification of high-risk situations, (3) identification of triggers, (4) stress level, (5) coping skills, and (5) quality of life. The text messages will include motivational messages and behavior-change techniques (e.g. coping with cravings and urges to drink, trigger identification, high-risk situation identification). Messages will encourage participants to continue with sobriety and focus on the success they have achieved so far.
  Other Names: Mobile Intervention
  Arms: Text Message (TM)

SUMMARY:
This is a research study of a text-messaging intervention to reduce alcohol relapse risk in pre-transplant liver transplantation patients. This study is an 8-week, randomized controlled pilot trial to investigate the feasibility and acceptability of a text-messaging intervention for alcohol relapse prevention and stress reduction in 20 liver transplant patients with alcohol-related liver disease. The goals of the study are (1) to develop a mobile, SMS-based stress reduction and alcohol use intervention for pre- liver transplant patients with alcohol-related liver disease (ALD) and (2) to evaluate the feasibility and acceptability of the mobile intervention and its effect on rates of alcohol consumption compared to a Standard Care condition in a liver transplantation center.

DETAILED DESCRIPTION:
This study is an 8-week, randomized controlled pilot trial to investigate the feasibility and acceptability of a text-messaging intervention for alcohol relapse prevention and stress reduction in 20 liver transplant patients with alcohol-related liver disease. The scientific aims of the study are as follows:

1. To develop a mobile, SMS-based stress reduction and alcohol use intervention for pre- liver transplant patients with alcohol-related liver disease (ALD).
2. Evaluate the feasibility and acceptability of the mobile intervention and its effect on rates of alcohol consumption compared to a Standard Care condition in a liver transplantation center.

Text messaging is a novel mechanism for intervention in this population. Over the course of the study, participants randomized to the Text Message condition will receive messages targeting known predictors of alcohol abstinence and relapse, including (1) craving, (2) identification of high-risk situations, (3) identification of triggers, (4) stress level, (5) coping skills, and (5) quality of life. Because mobile interventions have not been utilized in studies of alcohol abstinence, the protocol for this text message intervention on past studies that have used text messages interventions. Specifically, portions of a large-scale RCT of a text message intervention for smoking cessation and of a smaller study on a text message intervention for reducing alcohol-related consequences in college students. The text messages will include motivational messages and behavior-change techniques (e.g. coping with cravings and urges to drink, trigger identification, high-risk situation identification). Messages will encourage participants to continue with sobriety and focus on the success they have achieved so far. After the first 4 weeks, they will receive 3 messages per week for the next 4 weeks. All text messages will be developed with the input of liver transplant professionals.

All patients will be assessed at 4-weeks and 8-weeks and will provide urine for EtG analysis to allow biological verification of sobriety. After the 8-week intervention, patients will complete a satisfaction survey about their experiences in the Text Message condition and Standard Care condition to assess intervention helpfulness, text message content, and the ease of using the text message program. These data will allow the examination of the feasibility and acceptability of the text message intervention.

This study has two phases: (1) Stage 1 - development of intervention text messages and (2) Stage 2 - pilot randomized controlled trial of Text Message intervention versus Standard Care.

In Stage 1 - a text message bank of approximately 200-300 text messages will be developed using empirically supported in-person intervention components for heavy alcohol use and alcohol dependence. Component areas will be craving, high-risk situations, identification of alcohol use triggers, stress, mood, quality of life, and coping skills. As text messages will be used both for assessment and for intervention content, the text message bank will contain both assessment messages and intervention messages. Following the development of the text message bank, the messages will be assessed by Consultants to this project, which will include liver transplantation medical and psychological care providers. Text messages will be rated on their: (1) readability, (2) acceptability, (3) relevance to patients' concerns, and (4) helpfulness. Consultants will also be asked to indicate if they think any messages should be eliminated. Obtaining this feedback prior to the RCT will enhance the Text Message Intervention's acceptability to liver transplant providers.

Stage 2 is a between-subjects, randomized clinical trial that will compare the effect of a Text Message intervention with Standard Care in a liver transplantation clinic on alcohol relapse rate and stress reduction. This trial will also examine the feasibility and efficacy of the Text Message intervention. A total of 20 subjects, at least 18 years of age, will be recruited to participate in the trial and will be randomized to receive either the Text Message intervention or Standard Care. There are three consecutive phases to the study: (1) a 1-week assessment period; (2) an 8- week treatment period; (3) follow-up post-treatment and at 3-months post-intervention.

In Stage 2, we will conduct a randomized controlled pilot study to test the feasibility, acceptability, and preliminary efficacy of the final Text Message intervention versus a Standard Care (SC) intervention. Patients in the SC condition will receive all elements of their usual care as part of the liver transplant service but will not receive any text messages.

Screening: Participants who express interest in the study will attend an in-person intake to learn about the study, provide informed, voluntary consent, be further evaluated for eligibility and complete baseline assessments for which they will be compensated. Participants will be randomized to either the Text Message intervention or to SC based on a preset randomization schedule generated via computer by a statistician. For participants in the Text Message condition, the RA will demonstrate how to use the text messaging service. A pre-paid mobile phone will be provided for the duration of the study for all participants. Study cell phones will have pre-paid text messaging coverage for the duration of the study.

Interventions: In the SC condition, participants will receive only standard care provided by the liver transplantation team. No additional behavioral or psychosocial interventions will be provided. These participants will receive only study-specific assessments. Participants in this condition will complete assessments at baseline, 4-weeks and 8-weeks that measure self- reported substance use, stress, and coping skills. At each in-person assessment, participants will provide urine for EtG analysis.

In the Text Message condition, participants will receive daily text messages in addition to receiving all elements of standard care in the liver transplant service. Daily text messages will be used to determine their current level of functioning and provide text message intervention messages in response. Text messages will be sent via Google Voice on a research computer. A study-specific phone number will be generated via Google and will be the number from which all participants receive text messages. Participants will receive these messages on their pre-paid study cell phones only. Participants will be asked to respond to the text messages either with a specified response (e.g. YES/NO) or with a generic response (e.g. "1"). This will allow the collection of feasibility data on number of responses to the messages and verify that participants are reading and receiving the intervention. Participants' response messages will be received, via Google Voice, on a research computer. The research assistant will monitor and record whether a participant is responding at least once per day. As noted, some text messages will ask for a specific reply in response to a question (e.g. "Any cravings today?"). Based on the participant's response (e.g. "high," "med," or "low"), the research assistant will respond with a text message tailored to the participant's message. Participants will be informed that this account will be used for research purposes only and should not be used in the case of a clinical emergency, because all text messages have been pre-generated and it cannot be guaranteed that responses will be seen at the moment they are sent. All text messages will be sent to the HIC in an amendment to this protocol for approval.Over the course of the study, participants will receive messages targeting known predictors of alcohol abstinence and relapse, including (1) craving, (2) identification of high-risk situations, (3) identification of triggers, (4) stress level, (5) coping skills, and (5) quality of life. Because mobile interventions have not been utilized in studies of alcohol abstinence, we will base the protocol for this text message intervention on past studies that have used text message interventions. Specifically, we will apply portions a large-scale RCT of a text message intervention for smoking cessation and of a smaller study on a text message intervention for reducing alcohol-related consequences in college students. Following randomization, participants will receive 2 text messages per day for the first 4 weeks of the study. Research on the elaboration likelihood model of attitude change has indicated that tailored messages are more effective than generic messages. Because intervention messages are most effective if they are tailored to the personal characteristics of the participant, the daily text messages (content: craving, trigger identification, high-risk situation identification and other efficacious components of alcohol abstinence interventions) will be tailored on variables known to be risk factors for pretransplant abstinence, including gender, family history of alcoholism, and level of social support. The text messages will include motivational messages and behavior-change techniques (e.g. coping with cravings and urges to drink, trigger identification, high-risk situation identification). Messages will encourage participants to continue with sobriety and focus on the success they have achieved so far. After the first 4 weeks, they will receive 3 messages per week for the next 4 weeks. As noted, these messages will be developed with the input of liver transplant professionals. As in the Standard Care condition, participants in the Text Message condition will return to the liver clinic for assessments at 4-weeks and 8-weeks and to provide urine for EtG analysis.

End of Treatment Monitoring/Follow-Up: After the 8-week intervention, participants will be contacted via phone to schedule an in-person follow-up appointment. At follow-up participants will be asked to complete a satisfaction survey about their experiences with the Text Message or SC interventions. The survey will assess intervention helpfulness, text message content, and ease of using the text message program and will provide an end-of-treatment urine test.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* diagnosis of alcohol-related liver disease;
* currently in evaluation for UNOS listing as a liver transplant candidate;
* last reported use of any alcohol within the past 1 year;
* willingness to receive and respond to multiple text messages per day.

Exclusion Criteria:

* unstable psychiatric/medical conditions such as suicidal ideation, acute psychosis, or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2014-03-25 (Actual); Study Completion 2014-05-06 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility Evaluation | 8 weeks
  Patterns of text message usage
Alcohol Abstinence Rates | 8 Weeks
  Biologically confirmed (EtG) rates of abstinence from alcohol

SECONDARY OUTCOMES:
Subjective Alcohol Abstinence Rates | 8 Weeks
  Self-reports of any days drinking during treatment and self-reports of alcohol craving
Stress Ratings | 8 Weeks
  Perceived Stress Scale (PSS). Self-report 4 item scale with each item on a 0-4 scale (maximum score = 16). Higher scores indicate higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, PhD, Principal Investigator — Medical University of South Carolina; Kelly S DeMartini, PhD, Study Director — Yale Medical School
Locations (1):
- Yale Transplantation Center/Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Because the sample is so small, was collected at a very specific site with a specific sample, it could be possible for patients to be identified. Therefore, we have are not including data sharing.

REFERENCES:
- [Background] Free C, Knight R, Robertson S, Whittaker R, Edwards P, Zhou W, Rodgers A, Cairns J, Kenward MG, Roberts I. Smoking cessation support delivered via mobile phone text messaging (txt2stop): a single-blind, randomised trial. Lancet. 2011 Jul 2;378(9785):49-55. doi: 10.1016/S0140-6736(11)60701-0. PMID 21722952
- [Background] Weitzel JA, Bernhardt JM, Usdan S, Mays D, Glanz K. Using wireless handheld computers and tailored text messaging to reduce negative consequences of drinking alcohol. J Stud Alcohol Drugs. 2007 Jul;68(4):534-7. doi: 10.15288/jsad.2007.68.534. PMID 17568957
- [Background] Webb MS, Hendricks PS, Brandon TH. Expectancy priming of smoking cessation messages enhances the placebo effect of tailored interventions. Health Psychol. 2007 Sep;26(5):598-609. doi: 10.1037/0278-6133.26.5.598. PMID 17845111
- [Background] Pfitzmann R, Schwenzer J, Rayes N, Seehofer D, Neuhaus R, Nussler NC. Long-term survival and predictors of relapse after orthotopic liver transplantation for alcoholic liver disease. Liver Transpl. 2007 Feb;13(2):197-205. doi: 10.1002/lt.20934. PMID 17205563
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331

DOCUMENTS (2):
  • Informed Consent Form (2013-01-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT03402256/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2013-01-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT03402256/Prot_SAP_001.pdf